CLINICAL TRIAL: NCT05503823
Title: Investigating Transcranial Alternating Current Stimulation (tACS) Preconditioning Effects on Resting and Active Motor Threshold
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminary results indicate no significant difference in RMT pre- and post-tACS.
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HS25595 (B2022:070
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2022-08

CONDITIONS: Understand the Effects of tACS on the Brain
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: All participants will receive the same stimulations to analyze the effects of tACS on the brain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Participants (Experimental): Each participant will have their resting and active motor threshold measured using the transcranial magnetic stimulation (TMS) device. Participants will receive tACS for 10 minutes in the first session and tRNS in the second session.
  Interventions: Device: tACS or tRNS and TMS

INTERVENTIONS:
Device: tACS or tRNS and TMS — A light electrical current will be applied to the scalp of the participants via 2 electrodes. The resting and active motor threshold will be measured before, right after, after 30 minutes, and after 1 hour of receiving the tACS or tRNS.

SUMMARY:
Previous studies have looked at the potential of using transcranial direct current stimulation (tDCS) to prime the brain in order to lower the resting motor threshold. The resting motor threshold (RMT) is the intensity at which repeated transcranial magnetic stimulation (rTMS) is applied for treatments. The RMT is the lowest intensity at which the participant's muscle responds with the motor evoked potential peak-to-peak amplitude greater than 50μV for 5 of 10 trials when the hand is relaxed. The active motor threshold (AMT) is the lowest intensity that produces MEP with peak-to-peak amplitude greater than 100 μV for 5 of 10 trials while the participant maintains 10-30% of maximal voluntary contraction. The RMT and AMT is different for each person and the high intensity TMS pulses can be difficult for some of the patients in the current Alzheimer's rTMS treatment study to tolerate. Therefore, if the treatment can still be applied with lower intensities, it would be more tolerable for some people. The limited research on both tDCS and transcranial alternating current stimulation (tACS) in priming the brain for TMS are not enough to determine if they are effective in priming the brain. The studies that include tDCS have small sample size and inconclusive results. The studies with tACS are using very high frequencies of 140 Hz to 250 Hz. The objective of this research study is to determine if priming the brain with tACS at 40 Hz or tRNS for 10 minutes is able to reduce the resting and active motor threshold. Therefore, for people with higher RMT and AMT, priming with tACS or tRNS could be used to lower intensities while stimulating the brain for treatments.

DETAILED DESCRIPTION:
When volunteers are interested in participating in the study and they contact the PI or RA, the PI or RA will briefly explain the study. If the participant is still interested in participating, two 2-hour time slot will be scheduled for the participant to visit the lab. At the scheduled first visit, the PI or RA will provide and explain each part of the consent from. Once the participant is ready to participate, they will be asked to sign the consent form and will be provided a copy of the signed consent form. The PI or RA will assign a code to each participant. The code will be in the form of XY-RMT_##, where XY are the first letters of the first and last names and ## is a two digit number. After the consent form is signed, it will be placed in a locked cabinet located in our supervisor's office at Riverview Health Center.

Once the participant is fully enrolled, the RA and PI conduct the Montreal Cognitive Assessment (MoCA) and the Questionnaire to determine if the participant meets the inclusion criteria. If the participants have no health or physical conflicts with the application of electrical and magnetic stimulation and have a MoCA score higher than 26 out of 30, the PI and RA will set up the participant and the devices. Using our neuronavigation system in the TMS lab (at Riverview Health Center), a tracking headband will be placed on the participant and a tracker is used to measure the scalp and determine anatomical positions. Electrodes will also be placed on the participants first dorsal interosseous (FDI) muscle of the participant's right hand to record the electromyography (EMG).

The TMS device is the Magstim Rapid 2 Stimulator on single pulse setting with the figure-of-eight coil AirFilm Coil. The EMG device is the EMG Recording Pod from Brainsight 2. The tACS device is the Soterix Medical Inc. tES (transcranial electrical stimulation) (Model: 2001).

For the resting motor threshold (RMT), the PI exposes the participant's C3 section of the brain (area of the left hemisphere of the brain in 10 20 model which is related to the hand area of the primary motor cortex) to single pulses of TMS starting at 50% intensity of the maximum intensity available. This is done while the right hand is at a resting (relax) position. The RA will increase the intensity by increments of 5% until a visible twitch in the right hand is observed. Then the intensity will be decreased by decrements of 1% until 10 consistent visible twitches are observed in arrow. The minimum intensity is recorded as the RMT and the exact position and direction of the coil relative to the headband will be recorded as the target "hotspot" via the neuronavigational system (Vicra position sensor camera). The 10 consecutive successful EMGs will be recorded as the pre-priming data of the resting muscle. A similar procedure will be followed for the active motor threshold (AMT) with the only difference being the condition of the right hand. For an active recording, the participant will be asked to gently grab the arm rest of the chair so the muscle is activated 10-30% of maximal voluntary contraction and the 10 pulses will be exposed to the "hotspot as located by the Vicra camera.

To prime the brain using the tACS, the participant will be given a 5-minute break during which the RA places the active electrode of tACS on the marked "hotspot" and the reference on the contralateral supraorbital area of the head (right side of the forehead above the eyebrow). After the break, the stimulation begins at a frequency of 40 Hz and current intensity of 0.75 mA amplitude for duration of 10 minutes. Immediately after the stimulation the EMG will be recorded through 10 TMS pulses on active FDI muscle and 10 pulses with resting FDI muscle. The same procedure will be followed once 30 minutes after tACS stimulation and once after 1 hour. Similar procedure will be done for the right side RMT/AMT measurement which moves the left hand.

Overall, there will be 40 resting EMG recordings and 40 active EMG recording for each participant. The resting EMG recording will be compared at each time interval for any observable difference in average motor evoked potential (MEP) and the active EMG recordings are compared for difference in both the silence period which appears after the involuntary twitch and the MEP.

The same process will be done for a second time either 4 hours after the first session or on a different day. The only difference being that the participant receives 10 minutes of tRNS instead of tACS.

ELIGIBILITY:
Inclusion Criteria:

- Montreal Cognitive Assessment score greater than or equal to 26

Exclusion Criteria:

* being pregnant
* having any metallic implants in the head or upper body
* having a pacemaker
* having a history of seizures
* having a diagnosed major psychotic disorder
* having any nervous system medication (depression, anxiety, sleep, pain, etc.) on a daily basis
* having a brain injury

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Riverview Health Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Each participant will have their resting and active motor threshold measured using the transcranial magnetic stimulation (TMS) device. Participants will receive tACS for 10 minutes in the first session and tRNS in the second session.
  tACS or tRNS and TMS: A light electrical current will be applied to the scalp of the participants via 2 electrodes. The resting and active motor threshold will be measured before, right after, after 30 minutes, and after 1 hour of receiving the tACS or tRNS.
Period: Overall Study
Arm/Group | All Study Participants
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
MoCA score [Mean (Standard Deviation); unit: units on a scale] — Montreal Cognitive Assessment measures cognitive function with a maximum score of 30 and minimum score of 0. A score above 25 is considered normal. The lower the score means lower cognitive function.
  units on a scale | 27.9 (1.6)
Handedness [Count of Participants; unit: Participants]
  Right handed | 4
  Left handed | 2
Amount of sleep the night before [Mean (Standard Deviation); unit: hours] | 7.3 (1.1)
Anxiety [Median (Standard Deviation); unit: units on a scale] — Anxiety was determined on a scale from 1 to 5 where 1 represents no anxiety and 5 represents extremely anxious.
  units on a scale | 1.7 (0.5)
Pain medication [Count of Participants; unit: Participants]
  No | 6
  Yes | 0
Caffeine within 1 hour prior to study [Count of Participants; unit: Participants]
  No | 5
  Yes | 1

OUTCOME MEASURES:

1. Primary Outcome: Resting Motor Threshold
Description: The peak-to-peak amplitude of the muscle signal from the resting motor threshold.
Time Frame: Before tACS, right after tACS, 30 minutes after tACS, and 1 hour after tACS
Measure: Mean (Standard Deviation); unit: micro Volts
Groups:
- Resting Motor Threshold With tACS: Each participant will have their resting motor threshold measured using the transcranial magnetic stimulation (TMS) device. Participants will receive tACS for 10 minutes.
  tACS and TMS: A light electrical current will be applied to the scalp of the participants via 2 electrodes. The resting and active motor threshold will be measured before, right after, after 30 minutes, and after 1 hour of receiving the tACS or tRNS.
Arm/Group | Resting Motor Threshold With tACS
Number analyzed (Participants) | 6
micro Volts
  Before | 76.5 (26.6)
  After | 108.7 (43.2)
  30 min After | 130.1 (45)
  1 hour After | 85.8 (25.1)

2. Secondary Outcome: Active Motor Threshold
Description: Cortical silent period measured post-MEP.
Time Frame: Before tACS, right after tACS, 30 minutes after tACS, and 1 hour after tACS
Population: Majority of AMT data had significant noise, limiting the dataset to only 1 participant for all time frames.
Measure: Mean (Standard Deviation); unit: milli seconds
Groups:
- Active Motor Threshold With tACS: Each participant will have their resting motor threshold measured using the transcranial magnetic stimulation (TMS) device. Participants will receive tACS for 10 minutes.
  tACS and TMS: A light electrical current will be applied to the scalp of the participants via 2 electrodes. The resting and active motor threshold will be measured before, right after, after 30 minutes, and after 1 hour of receiving the tACS or tRNS.
Arm/Group | Active Motor Threshold With tACS
Number analyzed (Participants) | 1
milli seconds
  Before | 131.1
  After | 123.1
  30 min After | 81.4
  1 hour After | 108.75

ADVERSE EVENTS:
Time Frame: up to 4 hours
Description: Transcranial random noise stimulation (tRNS) was not tested due to lack of resources. We could not purchase the device that performed tRNS, therefore only tACS was performed for all study participants.
Groups:
- tACS Group; tRNS Group: Each participant will have their resting and active motor threshold measured using the transcranial magnetic stimulation (TMS) device.
  A light electrical current will be applied to the scalp of the participants via 2 electrodes. The resting and active motor threshold will be measured before, right after, after 30 minutes, and after 1 hour of receiving the tACS or tRNS.
Arm/Group | tACS Group | tRNS Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/0
Other Adverse Events (participants affected / at risk) | 0/6 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT05503823/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT05503823/ICF_001.pdf